CLINICAL TRIAL: NCT00826124
Title: Does MRI Improve Interventional Outcomes for Lumbosacral Radiculopathy? A Randomized Study Comparing Epidural Steroid Injections Based on Clinical Findings Alone, or Clinical Findings and MRI
Brief Title: Does Magnetic Resonance Imaging (MRI) Improve Interventional Outcomes for Lumbosacral Radiculopathy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Steven P. Cohen, MD, Johns Hopkins Medical Institutions, Pain Management Division
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00022479
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-01

CONDITIONS: Lumbosacral Radiculopathy
Keywords: low back pain; radiculopathy; sciatica
MeSH Terms: conditions — Low Back Pain; Radiculopathy; Sciatica | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Two epidural steroid injections two weeks apart based on history and physical exam alone
  Interventions: Procedure: Epidural steroid injection
- II (Active Comparator): Two epidural steroid injections two weeks apart based on history, physical exam and MRI
  Interventions: Procedure: Epidural steroid injection; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Epidural steroid injection — Injection based solely on history and physical exam
  Arms: I
Procedure: Epidural steroid injection — Two epidural steroid injections two weeks apart based on history, physical exam and MRI
  Arms: II
Procedure: Magnetic Resonance Imaging (MRI) — Imaging of lumbar spine
  Arms: II

SUMMARY:
Epidural steroid injections (ESI) are the most frequently performed procedures in pain clinics. When performing ESI, there is no consensus about how to best select candidates for this intervention, and which level(s) to inject. Some experts advocate basing the injection level on MRI findings, whereas others recommend clinical symptoms. In order to determine whether MRI is necessary before referring patients with chronic LBP radiating into the leg(s) for pain management interventions, we will perform a randomized comparative study involving 131 patients with chronic low back and leg pain who are clinically candidates for epidural steroid injections into two groups. Group I will receive two ESI based solely on historical and physical exam (PE) findings. Group II will receive treatment only after MRI is reviewed.

The investigators' hypothesis is that MRI will not have a significant effect on treatment outcome, and will have minimal impact on patient care.

DETAILED DESCRIPTION:
One hundred and thirty-one patients referred to the Blaustein Pain Treatment Center with back and leg pain will be randomized to receive one of two treatments. Sixty-three patients will be allocated to group I and up to 68 to group II (see below and statistical analysis). All patients will be candidates for ESI based on history and physical exam. All 63 group I patients will receive two ESI based solely on history and PE (i.e. the treating physician will be blinded to MRI results). Group II will receive treatment based on MRI, history and PE. This probably but may not include ESI (i.e. it is conceivable that a normal MRI might result in conventional therapy instead of ESI, though chemical irritation of nerve roots often occurs without disc protrusion. We estimate this to occur in no more than 10% of cases (probably less); hence, we are planning to randomize up to 68 patients to group II. If an ESI is done, the patient will receive two injections, similar to patients in group I. Randomization will be done by a research assistant via a computerized randomization system in groups of 13. In order to ensure no serious pathology is missed in group I subjects, a separate doctor with no knowledge of treatment allocation will review the films. If there is serious pathology such as evidence of spinal metastases or infection, the patient will be excluded from the study. There will be no "control" group in this study. Both evaluating physicians and patients will be blinded until they exit the study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Candidates for ESI based on history and physical exam
* NRS pain score > 4
* Leg pain > back pain
* Patients already have an MRI

Exclusion Criteria:

* Untreated coagulopathy
* Previous spine surgery
* Leg pain > 4 years duration
* Epidural steroid injection within past 2 years
* Serious (e.g., bowel or bladder incontinence, loss of reflexes) or progressive neurological deficit
* Referrals from surgery diagnostic injections for surgical evaluation
* Serious medical (e.g. congestive heart failure) or psychiatric (untreated depression) condition that might preclude optimal outcome
* Pregnancy
* Serious underlying pathology (e.g., vertebral fracture, spinal infection or metastases), as determined by an independent reviewer (group I) or the treating physician (group II) on MRI. The investigator and injector for group I patients will remain blinded to this review except to know that serious pathology was ruled out.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
change in numerical rating leg pain score | 1 month after 2nd epidural injection

SECONDARY OUTCOMES:
change in numerical rating back pain score | 1 month after 2nd epidural injection
change in numerical rating scale leg pain score | 3 months after 2nd epidural steroid injection
  Pain score 3 months after 2nd epidural steroid injection
Change in numerical rating scale back pain score | 3 months after 2nd epidural steroid injection
  Back pain 3 months after epidural steroid injections
Change in Oswestry disability index | 1 month after 2nd epidural steroid injection
  Measurement of functional capacity 1 month after 2nd epidural steroid injection
Change in Oswestry disability index | 3 months after 2nd epidural steroid injection
  Measurement of functional capacity 3 months after 2nd epidural steroid injection

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins School of Medicine, Baltimore, Maryland

REFERENCES:
- [Background] Kendrick D, Fielding K, Bentley E, Kerslake R, Miller P, Pringle M. Radiography of the lumbar spine in primary care patients with low back pain: randomised controlled trial. BMJ. 2001 Feb 17;322(7283):400-5. doi: 10.1136/bmj.322.7283.400. PMID 11179160
- [Background] Gilbert FJ, Grant AM, Gillan MG, Vale LD, Campbell MK, Scott NW, Knight DJ, Wardlaw D; Scottish Back Trial Group. Low back pain: influence of early MR imaging or CT on treatment and outcome--multicenter randomized trial. Radiology. 2004 May;231(2):343-51. doi: 10.1148/radiol.2312030886. Epub 2004 Mar 18. PMID 15031430
- [Background] Modic MT, Obuchowski NA, Ross JS, Brant-Zawadzki MN, Grooff PN, Mazanec DJ, Benzel EC. Acute low back pain and radiculopathy: MR imaging findings and their prognostic role and effect on outcome. Radiology. 2005 Nov;237(2):597-604. doi: 10.1148/radiol.2372041509. PMID 16244269
- [Background] Cohen SP, Argoff CE, Carragee EJ. Management of low back pain. BMJ. 2008 Dec 22;337:a2718. doi: 10.1136/bmj.a2718. No abstract available. PMID 19103627
- [Derived] Cohen SP, Gupta A, Strassels SA, Christo PJ, Erdek MA, Griffith SR, Kurihara C, Buckenmaier CC 3rd, Cornblath D, Vu TN. Effect of MRI on treatment results or decision making in patients with lumbosacral radiculopathy referred for epidural steroid injections: a multicenter, randomized controlled trial. Arch Intern Med. 2012 Jan 23;172(2):134-42. doi: 10.1001/archinternmed.2011.593. Epub 2011 Dec 12. PMID 22157067